CLINICAL TRIAL: NCT05853458
Title: HU-F-AIM - A Prospective, Interventional Study to Evaluate HU-resistance in Polycythemia Vera Patients Who Meet Predictive Parameters Identified in the Machine Learning Project PV-AIM
Brief Title: Evaluation of HU-resistance in Adult Patients With Polycythemia Vera Who Meet PV-AIM Predictors
Acronym: HU-F-AIM
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424BDE15; 2022-502338-20-00 (Other: EU CTIS number)
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Polycythemia Vera
Keywords: Polycythemia vera (PV); Hydroxyurea; Resistance; Intolerance; Predictive parameters
MeSH Terms: conditions — Polycythemia Vera | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydroxyurea (HU) (Experimental): Participants will be treated with HU capsules, orally taken, for a maximum duration of 15 months.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — Hydroxyurea is commercially available in Germany and will be prescribed based on clinical judgment

SUMMARY:
The purpose of this study is to confirm the predictive factors for hydroxyurea (HU) failure (hemoglobin (HGB) <15.5 g/dL (9.62 mmol/L) and red blood cell distribution width (RDW) ≥17%) identified by machine learning in the polycythemia vera advanced integrated model (PV-AIM) project in the real-life setting.

DETAILED DESCRIPTION:
The study consists of three periods: Screening period, treatment period (observation for HU-resistance/intolerance) and follow-up (FU) period.

Eligible participants will enter the treatment period (observation period for HU-resistance/intolerance) and start receiving the de novo HU treatment. The maximum treatment duration for each participant in the study will be up to 15 months.

This study will be conducted in a total of 300 adult PV patients and approximately at 30 to 40 sites in Germany. If necessary, the study will be extended to other countries to achieve the target population.

ELIGIBILITY:
Key Inclusion criteria

1. Signed informed consent must be obtained prior to participation in the study
2. Patients ≥18 years
3. Confirmed diagnosis of Polycythemia vera (according to WHO 2008, 2016, or 2022 criteria) (Tefferi and Vardiman 2008, Arber et al 2016, Khoury et al 2022)
4. Eastern Cooperative Oncology Group (ECOG) ≤ 2
5. No previous pharmacologic cytoreductive therapy (including investigational drugs)
6. No phlebotomy in last 14 days
7. HU-eligible

   * High-risk: age ≥ 60 years and/or prior history of thrombosis
   * Low-risk: showing at least one of the defined criteria

     * Signs of disease progression (myeloproliferation):

       * Increase in spleen size or symptomatic splenomegaly
       * Platelet increase to > 1,000,000/µl
       * WBC increase to > 15,000/µl or higher
       * Frequent (> 10 per year) or increasing frequency of phlebotomies
     * Increasing risk of thromboembolism and bleeding:

       * New thromboembolism and/or hemorrhagic complications
       * Microcirculation disorders despite acetyl salicylic acid (ASA) 2x 100 mg/day
       * Restricted feasibility or intolerance of phlebotomies
       * Symptomatic iron deficiency
       * Uncontrolled increase in hematocrit
       * Severe or distressing disease-related symptoms
8. Female participants of childbearing potential should have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study treatment.

Key Exclusion criteria

1. Patients with post-polycythemia vera myelofibrosis (post-PV MF) or accelerated phase/ blast phase myeloproliferative neoplasm acute myeloid leukemia (AP/BP-MPN AML).
2. Patients with a contraindication to HU according to the SmPC (severe bone marrow depression, leukopenia (< 2.5 x 109 leukocytes/l), thrombocytopenia (< 100 x 109 platelets/L), severe anemia (< 10 g/dL HGB).
3. Patients with rare hereditary galactose intolerance, total lactase deficiency or glucose-galactose malabsorption in their past medical history.
4. Active uncontrolled infection that is considered by the Investigator as a reason for exclusion.
5. Active malignancies (except for carcinoma in situ; prostate cancer and breast cancer in remission and - where necessary - ongoing hormonal therapy).
6. Inadequate renal function as demonstrated by Modification of Diet in Renal Disease estimate glomerular filtration rate (MDRDeGFR) < 30 mL/min/1.73m2 or on dialysis.
7. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotrophin (hCG) laboratory test.
8. Sexually active males unwilling to use a condom during intercourse while taking study treatment and for at least 3 months after stopping study treatment.
9. HIV patients treated with nucleoside reverse transcriptase inhibitors like didanosine and stavudine.

Other inclusion/exclusion criteria may apply

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2027-01-27 (Estimated); Study Completion 2027-01-27 (Estimated)

PRIMARY OUTCOMES:
Proportion of PV patients with HU-resistance/intolerance within 6-9 months after start of de novo HU- treatment in presence of the PV-AIM HU-resistance predictors at the start of HU treatment. | From 6 to 9 months after start of de novo HU-treatment
  Proportion of PV participants with HU resistance/intolerance within 6-9 months after start of de novo HU treatment in presence of the PV-AIM HU resistance predictors at the start of HU treatment. The proportion will be assessed calculating the rate together with the respective 95% confidence interval (CI).

SECONDARY OUTCOMES:
Proportion of PV patients who meet the PV-AIM HU-resistance predictors before start of HU-treatment | Baseline
  Proportion of PV patients who meet the PV-AIM HU-resistance predictors before start of HU-treatment. The proportion will be assessed calculating the rate together with the respective 95% confidence interval (CI).
Proportion of patients developing HU resistance/intolerance at any time within the maximum treatment period of 15 months | Up to 15 months
  Proportion of patients developing HU resistance/intolerance at any time within the maximum treatment period of 15 months. The proportion will be assessed calculating the rate together with the respective 95% confidence interval (CI).
Proportion of "non-switchers" | Up to 15 months
  For all patients who develop HU resistance/intolerance according to modified European LeukemiaNet (ELN) criteria at any time during the maximum treatment period of 15 months, the proportion of "non-switchers" (i.e., patients remaining on HU despite they meet the HU-resistance/intolerance criteria) will be assessed. The rate will be calculated together with the respective 95% confidence interval (CI).
Timepoint of therapy switch (after confirmation of HU resistance/intolerance) | Up to 15 months
  For all patients who develop HU resistance/intolerance according to modified ELN criteria at any time during the maximum treatment period of 15 months, the timepoint of therapy switch (after confirmation of HU resistance/intolerance) will be assessed.
Reasons for therapy switch / non-switch | Up to 15 months
  For all patients who develop HU resistance/intolerance according to modified ELN criteria at any time during the maximum treatment period of 15 months, the reasons for therapy switch or non-switch will be summarized
Therapies applied during follow-up period | Up to 3 months after treatment discontinuation
  For all patients who develop HU resistance/intolerance according to modified ELN criteria at any time during the maximum treatment period of 15 months, the therapies applied during the follow-up period will be summarized

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- Germany (23):
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Kronach, Bavaria
  - Novartis Investigative Site, Straubing, Bavaria
  - Novartis Investigative Site, Langen, Hesse
  - Novartis Investigative Site, Lingen Ems, Lower Saxony
  - Novartis Investigative Site, Aachen, North Rhine-Westphalia
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Dortmund, North Rhine-Westphalia
  - Novartis Investigative Site, Velbert, North Rhine-Westphalia
  - Novartis Investigative Site, Saarbrücken, Saarland
  - Novartis Investigative Site, Merseburg, Saxony-Anhalt
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Donauwörth
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erding
  - Novartis Investigative Site, Gütersloh
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Mutlangen
  - Novartis Investigative Site, Naunhof
  - Novartis Investigative Site, Westerstede
  - Novartis Investigative Site, Würselen

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com